CLINICAL TRIAL: NCT02131103
Title: The Short- and Long Term Outcomes of Early Routine PCI With the Standard Treatment in Low-intermediate Risk ST-elevation Myocardial Infarction Patients Who Successfully Fibrinolysis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Yotsawee Chotechuang, Chiang Mai University, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COM-2556-01631
Record Dates: First submitted 2014-05-03; First posted 2014-05-06 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2014-05

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Pharmacoinvasive strategy
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Early ( < 24hr) (Active Comparator): Early percutaneous coronary intervention means performed coronary intervention between 3-24 hours after successful fibrinolytic therapy.
  Interventions: Other: Percutaneous coronary intervention
- Delay ( > 24 hours) (Active Comparator): Delay percutaneous coronary intervention means received coronary intervention >24 hours to 2 weeks after successfully fibrinolytic therapy.
  Interventions: Other: Percutaneous coronary intervention
- Early (Active Comparator): We randomized the patients into two groups early (≤ 24 hours) and delay group (> 24 hours) All patients received fibrinolysis, aspirin 300 mg and clopidogrel (300 mg for participants 75 years of age or younger or 75 mg for participants older than 75 years of age). Patients older than 75 years of age did not receive enoxaparin.
  Patients will be randomly assigned to either the group that received routine early PCI (hereinafter termed the early-PCI group) or the group that received standard treatment (PCI performed after 24-72 hours of successfully fibrinolysis). Randomized will perform within 24 hours after successful fibrinolytic therapy. PCI will be performed when persistent occlusion or substantial stenosis of the infarct-related artery (either stenosis of 70% or more of the diameter of the artery or stenosis of 50-70% with thrombus, ulceration, or spontaneous dissection) was present. In case of multivessel disease, only culprit lesion will be correct.
  Interventions: Other: Percutaneous coronary intervention

INTERVENTIONS:
Other: Percutaneous coronary intervention — All patients received fibrinolysis, aspirin 300 mg and clopidogrel (300 mg for participants 75 years of age or younger or 75 mg for participants older than 75 years of age). Patients older than 75 years of age did not receive enoxaparin.
  Patients will be randomly assigned to either the group that received routine early PCI (hereinafter termed the early-PCI group) or the group that received standard treatment (PCI performed after 24-72 hours of successfully fibrinolysis). Randomized will perform within 24 hours after successful fibrinolytic therapy. PCI will be performed when persistent occlusion or substantial stenosis of the infarct-related artery (either stenosis of 70% or more of the diameter of the artery or stenosis of 50-70% with thrombus, ulceration, or spontaneous dissection) was present. In case of multivessel disease, only culprit lesion will be correct.

SUMMARY:
1. Objective: To evaluate short- and long-term in the STEMI patients who successfully thrombolysis with early routine and delay percutaneous coronary intervention in low-intermediate risk patients.
2. Educational/ application advantages: To evaluate the time of early and delay PCI after received fibrinolysis had an effect to the short- and long-term clinical outcomes in low- intermediate GRACE risk score patients. No available of randomized controlled study in these group of the patients.

DETAILED DESCRIPTION:
1.Research design: Intervention trial 1.1 Study domain: STEMI patients who will receive the fibrinolysis for reperfusion therapy 1.2 Target population: STEMI patients who will receive the percutaneous coronary intervention after fibrinolysis in Lampang Regional hospital and Maharaj Nakorn Chiang Mai hospital.

1.3 Study population: STEMI patients who will receive the percutaneous coronary intervention after fibrinolysis during the year of 2013-2014 at Lampang Regional hospital and Maharaj Nakorn Chiang Mai hospital

Inclusion criteria:

1. The patients who received the percutaneous coronary intervention after fibrinolysis
2. Adult patients with age more than 18 years old
3. GRACE risk score less than 155 (low-intermediate risk)

Exclusion criteria:

1. The patients who received primary PCI or rescue PCI
2. The patients who had the previous history of coronary-artery bypass surgery
3. The high risk patients (such as cardiogenic shock, complete heart block, GRACE ≥155)

1.4 Occurrence relation Y (Composite outcomes) = f (Treatment early vs. delay | confounders)

1.5 Setting: The study will be conducted in Lampang Regional hospital and Maharaj Nakorn Chiang Mai hospital.

1.6 Determinant (x): Time to percutaneous coronary intervention (early vs. delayed).

1.7 Events (y): composite outcomes (included of death, re-infarction, and recurrent ischemia), re-hospitalized with ACS, and worsening heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. The patients who received the percutaneous coronary intervention after fibrinolysis
2. Adult patients with age more than 18 years old
3. GRACE risk score less than 155 (low-intermediate risk)

Exclusion Criteria:

1. The patients who received primary PCI or rescue PCI
2. The patients who had the previous history of coronary-artery bypass surgery
3. The high risk patients (such as cardiogenic shock, complete heart block, GRACE ≥155)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
composite outcomes(included of death, re-infarction, and recurrent ischemia), re-hospitalized with ACS, and worsening heart failure. | 6 months
  Composite outcomes included of death, re-infarction, recurrent ischemia, re-hospitalized with ACS and worsening heart failure at 30 days for short- and 6 months for long-term outcomes.
  Death was defined as all cause of death (cardiac and non-cardiac cause). Recurrent MI 'Incident MI' is defined as the individual's first MI. Re-infarction The term of 're-infarction' is used for an acute MI that occurs within 28 days of an incident- or recurrent MI.
  Re-hospitalized with ACS was defined as re-admission after discharge from hospital with acute coronary syndrome composed with clinical chest pain, rising of cardiac enzymes and dynamic ST-segment change.
  Re-hospitalized with heart failure was defined as re-admission after discharge from hospital with clinical decompensated heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Chiang Mai University, Chiang Mai, Chiang Mai, Thailand

REFERENCES:
- [Derived] Chotechuang Y, Phrommintikul A, Kuanprasert S, Muenpa R, Patumanond J, Chaichuen T, Sukonthasarn A. Cardiovascular outcomes of early versus delayed coronary intervention in low to intermediate-risk patients with STEMI in Thailand: a randomised trial. Heart Asia. 2019 Jun 12;11(2):e011201. doi: 10.1136/heartasia-2019-011201. eCollection 2019. PMID 31275432